CLINICAL TRIAL: NCT05515419
Title: Allogeneic Cord Blood in the Treatment of Neurological Diseases in Adults
Brief Title: Allogeneic Cord Blood for Neurological Diseases in Adults
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to regulatory reasons
Sponsor: The Medical Pavilion Bahamas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neurological Diseases; Stroke; Spinal Cord Injuries
Keywords: Adults
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: allogeneic cord blood for adult patients with neurological diseases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic cord blood therapy (Experimental): Allogeneic cord blood therapy
  Interventions: Biological: Allogeneic cord blood treatment

INTERVENTIONS:
Biological: Allogeneic cord blood treatment — Allogeneic cord blood treatment

SUMMARY:
This open label trial is conducted to investigate the efficacy and safety of allogeneic umbilical cord blood therapy for adult patients with neurological diseases.

DETAILED DESCRIPTION:
Neurological diseases such as stroke or spinal cord injuries are very common etiologies causing disability in developed countries. Cord blood possess various stem and progenitor cells, as well as their secreted regenerative factors, and is known to repair injured brain. The investigators clinical research aims to determine the safety and efficacy of allogeneic Umbilical Cord Blood for adult patients with neurological diseases such as stroke and spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke (onset < 24 months), or
* Spinal cord injury (onset < 24 months)

Exclusion Criteria:

* Raised intracranial pressure
* Malignant cancer
* Renal failure
* Severe pulmonary dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in modified Rankin Scale (mRS) | 1 month - 3 months - 6 months - 12 months
  modified Rankin Scale (mRS) from 1 - 5 whereby 1 is best (no significant disability) and 5 is worst (severe disability); The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.

SECONDARY OUTCOMES:
Monitoring Adverse Events | 1 month - 3 months - 6 months - 12 months
  Number of participants with treatment-related adverse events as assessedCommon by Toxicity Criteria for Adverse Events (CTCAE).version 5.0; adverse events are graded on a scale from 0 to 5, whereby grade 0 is best (no AE) and grade 5 is worst (fatal).

CONTACTS AND LOCATIONS:
Overall Officials: Conville S Brown, MD, Principal Investigator — The Medical Pavilion Bahamas

IPD SHARING:
Plan to Share IPD: No